CLINICAL TRIAL: NCT03758235
Title: Incobotulinumtoxin Versus Onabotulinumtoxin in the Treatment of Patients With Overactive Bladder Syndrome
Brief Title: Overactive Bladder Syndrome: Incobotulinumtoxin Versus Onabotulinumtoxin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Antonella Giannantoni, PA, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Inco_Ona
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Overactive Bladder Syndrome
Keywords: overactive bladder syndrome; botulinum toxin type A; onabotulinumtoxin/A; incobotulinumtoxin/A; treatment; neurogenic detrusor overactivity incontinence; urinary incontinence; urinary tract infections
MeSH Terms: conditions — Urinary Incontinence; Urinary Tract Infections | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the 4 groups (Incobot/A Group different dosages, or Onabot/A Group different dosages ) in parallel for the duration of the study.
Who Masked: Participant, Investigator
Masking Description: Partecipants, investigators and outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Incobot/A 100 U (Experimental): Incobot/A 100 U diluted in 10 ml of sodium chloride solution 0.9% by endoscopic detrusor injections (20 injections, 0.5 ml of solution for each injection) will be administered in patients able to perform spontaneous micturitions
  Interventions: Drug: IncobotulinumtoxinA 100 UNT Injection [Xeomin]
- Incobot/A 200 U (Experimental): Incobot/A 200 U diluted in 30 ml of sodium chloride solution 0.9% by endoscopic detrusor injections (30 injections, 1 ml of solution for each injection) will be administered in patients performin intermittent catheterization.
  Interventions: Drug: IncobotulinumtoxinA 100 UNT Injection [Xeomin]
- Onabot/A 100 U (Active Comparator): Onabot/A 100 U diluted in 10 ml of sodium chloride solution 0.9% by endoscopic detrusor injections (20 injections, 0.5 ml of solution for each injection) will be administered in patients able to perform spontaneous micturitions
  Interventions: Drug: OnabotulinumtoxinA 100 UNT [Botox]
- Onabot/A 200 U (Active Comparator): Onabot/A 200 U diluted in 30 ml of sodium chloride solution 0.9% by endoscopic detrusor injections (30 injections, 1 ml of solution for each injection) will be administered to patients performing intermittent catheterization
  Interventions: Drug: OnabotulinumtoxinA 100 UNT [Botox]

INTERVENTIONS:
Drug: IncobotulinumtoxinA 100 UNT Injection [Xeomin] — Incobot/A intradetrusor injections under cystscopic guidance, with local anaethesia in an outpatient basis
  Other Names: Incobot/A
  Arms: Incobot/A 100 U; Incobot/A 200 U
Drug: OnabotulinumtoxinA 100 UNT [Botox] — Onabot/A intradetrusor injections under cystscopic guidance, with local anaethesia in an outpatient basis
  Other Names: Onabot/A
  Arms: Onabot/A 100 U; Onabot/A 200 U

SUMMARY:
The aim of the original study was to compare Incobot/A versus Onabot/A in order to evaluate if the differences in the pharmacologic formulations between the two drugs could affect their efficacy and safety in the treatment of neurogenic overactive bladder (OAB).

In the original study protocol two different dosages for either Incobot/A and Onabot/A (200 U and 100 U) were considered, to treat patients with neurogenic detrusor overactivity incontinence performing intermittent catheterization (IC) with higher dosages and those able to void spontaneously with lower dosage, with the resulting four treatment groups. For such a study, a very large sample of participants should have been treated and followed up, to have adequate power to demonstrate the hypothesis. At the end of last February 2020, we had to temporarily stop all the clinical activities related to the study and patients' recruitment, due to the occurrence of Sars-Cov-2 pandemic in our Country. At that point, a non-inferiority study seemed to be possible and adequate, and we adapted the protocol accordingly. In addition, on the basis of previously published information, we could hypothesize that the new drug (Incobot/A) would have had at least a roughly similar effect to the control drug (Onabot/A). In order to perform a non-inferiority study, the power and sample size analysis have been re-planned.

Thus, we perform a not planned interim analysis to show the preliminary results of an ongoing, non-inferiority trial in which patients' recruitment temporarily stopped due to incontrollable external factors. The present study will be aimed to assess the non-inferiority of Incobot/A compared to Onabot/A on the efficacy and safety parameters, in the treatment of patients with refractory NDOI performing IC, who are randomized to receive 200 U of Incobot/A or Onabot/A intradetrusor injections and who are followed up to 12 wks after treatment

DETAILED DESCRIPTION:
This is a pilot, prospective, randomized, double blinded, multicentre, clinical trial. After giving a written informed consent, all the patients will be randomized into two groups: Group 1, including patients who will be treated with the Incobot/A and Group 2, including patients who will be treated with Onabot/A. The randomization process will be made by a computerized system. Enrolling period: September 2018- April 2020.

Inclusion criteria:

* patients (males and females) with neurogenic urge urinary incontinence (UUI) (with urgency, increase in day- time and night- time urinary frequency) and with urodynamic diagnosis of detrusor overactivity (DO);
* 18- 80 years;
* women of childbearing age, who use a reliable method of contraception throughout the study period (a pregnancy test must be performed during enrolment in the study);
* spinal cord injury at or below T1, diagnosed at least 6 months before the screening in case of a vesico-sphincter dysfunction due to spinal cord injury;
* EDSS score ≤ 6, in MS patients;
* patients refractory to anticholinergic therapy (≥ 1 anticholinergic agent)
* application of intermittent catheterizations to empty the bladder. In the case of spontaneous micturition, the patients should agree for the use of intermittent catheterizations, in case this will be necessary after treatment with the detrusor injection of botulinumtoxin A.

Urodynamic characteristics:

urodynamic diagnosis of DO, refractory to standard anticholinergics and naïve to intradetrusor injection of onabotulinumtoxin A.

The wash- out period after anticholinergics should be of at least 3 weeks. It will be also possible for patients continuing to assume previous anticholinergic therapy through the study period.

Exclusion criteria:

* recurring urinary tract infections (UTIs) (≥ 4 episodes/year);
* spinal cord injuries above T1;
* MS patients: EDSS score ≥ 6;
* patients who won't or can't perform intermittent catheterization;
* pregnancy or breast- feeding, if female patients
* post- void residual volume (PRV) > 150 ml, in the case of spontaneous micturition

Time 0 (pre-screening):

* history and physical examination;
* urinalysis and cultures (pregnancy test);
* 3- days voiding diary;
* urodynamic study;
* "Incontinence Quality of Life" (I- QoL) standardized Questionnaire;
* Visual Analog Scale (VAS) for evaluation of treatment satisfaction.

Time 1. Treatment.

Patients will be randomized into two groups, assigned by a computerized system:

- Group 1- Incobot/A:

patients with spontaneous micturitions will undergo only one administration of Incobot/A 100 U diluted in 10 ml of sodium chloride solution 0.9% by endoscopic detrusor injections (20 injections, 0.5 ml of solution for each injection); patients who perform intermittent catheterization will undergo only one administration of Incobot/A 200 U diluted in 30 ml of sodium chloride solution 0.9% by endoscopic detrusor injections (30 injections, 1 ml of solution for each injection)

- Group 2- Onabot/A:

patients with spontaneous micturitions will undergo only one administration of Onabot/A 100 U diluted in 10 ml of sodium chloride solution 0.9% by endoscopic detrusor injections (20 injections, 0.5 ml of solution for each injection); patients who perform intermittent catheterization will undergo only one administration of Onabot/A 200 U diluted in 30 ml of sodium chloride solution 0.9% by endoscopic detrusor injections (30 injections, 1 ml of solution for each injection)

Follow-up:

History and physical examination, 3-day voiding diary and VAS were repeated at 2, 4 and 12 weeks, in order to make better comparisons with previously published pivotal trials on Botox. Urinalyses and cultures and I-QoL questionnaire were repeated at 2 and 12 weeks after treatment; urodynamic examination was obtained at 12 weeks follow- up.

Outcomes of the study The primary outcome measure is change from baseline in the daily frequency of UI at week 12. Secondary outcomes measures are: the occurrence of UTIs and other treatment-related local and systemic adverse events following the two botulinum toxins A injections, during the observation period; changes from baseline in I-QOL total score and VAS scores (week 2 and week 12); changes from baseline in MCC, first volume and maximum pressure of detrusor overactivity (weeks 12), following the two botulinum toxins A administration.

Statistical Analysis:

In a non- inferiority trial, it is recommended to set the non-inferiority limit below the minimal clinically important difference such that, after the intervention, the two groups are expected to differ by less than this difference. Group sample sizes of 50 and 50 subjects are required to be 80% sure that the higher limit of 95% confidence interval was below the clinically important non-inferiority limit of + one in UI episodes/day between the experimental and the standard treatment. The true difference between the means is assumed to be 0 with standard deviation (SD) of 2. The significance level (alpha) of the test is 0.05. The sample size is calculated using PASS 11.0.7, Power Analysis and Sample Size Software (2011). NCSS, LLC. Kaysville, Utah, USA. In establishing the non-inferiority margin, we have considered one incontinence episodes/day as non-inferiority limit as the difference of one less urinary incontinence episode represents the smallest difference that can be measured in the count. Moreover, when considering the frequency of daily urinary incontinence (UI) at baseline in both groups of treatment, one UI episode represents about 15%. In the present study, due to the temporary stop of patients' recruitment, a not planned interim analysis of the current data from the ongoing trial is conducted, in order to detect whether the research outcomes will be addressed. The true difference between the means is assumed to be 0 with SD of 2. The significance level (alpha) of the test is 0.05. The sample size is calculated using PASS 11.0.7, Power Analysis and Sample Size Software (2011). NCSS, LLC. Kaysville, Utah, USA. The primary endpoint was analysed using a standard analysis of covariance (ANCOVA) model, including treatment group as fixed factors and baseline UI episodes/day as a covariate. If the higher one-sided 95% confidence interval (CI) limit that is produced from the ANCOVA model is lower than + one UI episode, the efficacy of the experimental treatment group is considered not inferior to that of the standard treatment group. Mann-Whitney's U-test is used for comparisons of unpaired data and Friedman and Wilcoxon tests for comparisons of paired data, X2 with Yates' continuity correction or Fisher's exact test are used to analyse categorical data. All statistical analyses are performed using IBM-SPSS® version 26.0 (IBM Corp., Armonk, NY, USA, 2019). In all analyses, a two-sided p-value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patients (males and females) with neurogenic urge urinary incontinence (UUI) (with urgency, increase in day- time and night- time urinary frequency) and with urodynamic diagnosis of DO;
* 18- 80 years;
* women of childbearing age, who use a reliable method of contraception throughout the study period (a pregnancy test must be performed during enrolment in the study);
* spinal cord injury at or below T1, diagnosed at least 6 months before the screening in case of a vesico-sphincter dysfunction due to spinal cord injury;
* EDSS score ≤ 6, in MS patients;
* patients refractory to anticholinergic therapy (≥ 1 anticholinergic agent)
* application of intermittent catheterizations to empty the bladder. In the case of spontaneous micturition, the patients should agree for the use of intermittent catheterizations, in case this will be necessary after treatment with the detrusor injection of botulinumtoxin A.

Exclusion Criteria:

* recurring urinary tract infections (UTIs) (≥ 4 episodes/year);
* spinal cord injuries above T1;
* MS patients: EDSS score ≥ 6;
* patients who won't or can't perform intermittent catheterization;
* pregnancy or breast- feeding, if female patients;
* post- void residual volume (PRV) > 150 ml, in the case of spontaneous micturition;
* hypersensitivity to the active substance or to any of the excipients (listed in section 6.1 of RCP);
* generalized diseases of muscular activity (e.g. myasthenia gravis, Lambert-Eaton syndrome);
* presence of infection or inflammation at the injection site;
* patients with acute urinary retention at the time of treatment, not routinely subjected to catheterization;
* men with overactive bladder and signs or symptoms of urinary obstruction should not be treated;
* documented or suspected active malignant neoplasia or previous history, within 2 years prior to screening;
* patients who must or want to continue taking illegal drugs or drugs that may interfere with the proper conduct of the study;
* chronic abuse of alcohol or drugs or any condition that in the opinion of the investigator doctor makes an unreliable subject in correctly completing the study procedures;
* any other clinical condition that would endanger the safety of patients in participating in the study or that could prevent the subjects from adhering to the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the frequency of urinary incontinence episodes. | 24 weeks
  change from baseline in the daily frequency of urinary incontinence episodes, as assessed by the 3-day voiding diary.
Evaluation of frequency of urinary tract infections in both arms of treatment. | 2, 12, 24 weeks
  Measurement of eventual differencies between the two arms of treatment in the frequency of urinary tract infections at 2, 12 and 24 weeks after treatment

SECONDARY OUTCOMES:
Change from baseline in urodynamic parameters. | 24 weeks
  Significant improvements in urodynamic parameters (maximum cystometric capacity, maximum detrusor pressure during first involuntary detrusor contraction) at 12 and 24 weeks as compared to baseline.
Change from baseline in Incontinence Quality of Life (I-QoL) questionnaire total score. | 2, 12, 24 weeks
  Significant improvement in I-QoL total score at 2, 12 and 24 weeks as compared to baseline.
Recording of the adverse events. | 2, 12, 24 weeks
  Assessment of possible adverse events-AE (systemic AEs: fatigue, weakness, dyspnoea, gastrointestinal irritation, Flu-like symptoms, dizziness; local AEs: haematuria, dysuria, urinary retention, post-void residual volume > 150 ml) at 2, 12 and 24 weeks after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Giannantoni, M.D., Principal Investigator — University of Siena; Emanuele Rubilotta, MD, Study Chair — Universita di Verona; Matteo Balzarro, MD, Study Director — Universita di Verona
Locations (1):
- Antonella Giannantoni, Siena, SI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohee A, Khan A, Harris N, Eardley I. Long-term outcome of the use of intravesical botulinum toxin for the treatment of overactive bladder (OAB). BJU Int. 2013 Jan;111(1):106-13. doi: 10.1111/j.1464-410X.2012.11282.x. Epub 2012 Jun 6. PMID 22672569
- [Result] Thuroff JW, Abrams P, Andersson KE, Artibani W, Chapple CR, Drake MJ, Hampel C, Neisius A, Schroder A, Tubaro A. EAU guidelines on urinary incontinence. Eur Urol. 2011 Mar;59(3):387-400. doi: 10.1016/j.eururo.2010.11.021. Epub 2010 Nov 24. PMID 21130559
- [Result] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Lemack GE, Dewey RB Jr, Roehrborn CG, O'Suilleabhain PE, Zimmern PE. Questionnaire-based assessment of bladder dysfunction in patients with mild to moderate Parkinson's disease. Urology. 2000 Aug 1;56(2):250-4. doi: 10.1016/s0090-4295(00)00641-5. PMID 10925088
- [Result] Aharony SM, Lam O, Corcos J. Evaluation of lower urinary tract symptoms in multiple sclerosis patients: Review of the literature and current guidelines. Can Urol Assoc J. 2017 Jan-Feb;11(1-2):61-64. doi: 10.5489/cuaj.4058. PMID 28443147
- [Result] Wyndaele JJ. The management of neurogenic lower urinary tract dysfunction after spinal cord injury. Nat Rev Urol. 2016 Dec;13(12):705-714. doi: 10.1038/nrurol.2016.206. Epub 2016 Oct 25. PMID 27779229
- [Result] Campos-Sousa RN, Quagliato E, da Silva BB, de Carvalho RM Jr, Ribeiro SC, de Carvalho DF. Urinary symptoms in Parkinson's disease: prevalence and associated factors. Arq Neuropsiquiatr. 2003 Jun;61(2B):359-63. doi: 10.1590/s0004-282x2003000300007. Epub 2003 Jul 28. PMID 12894267
- [Result] Kanai A, Andersson KE. Bladder afferent signaling: recent findings. J Urol. 2010 Apr;183(4):1288-95. doi: 10.1016/j.juro.2009.12.060. Epub 2010 Feb 19. PMID 20171668
- [Result] Veenboer PW, Bosch JL. Long-term adherence to antimuscarinic therapy in everyday practice: a systematic review. J Urol. 2014 Apr;191(4):1003-8. doi: 10.1016/j.juro.2013.10.046. Epub 2013 Oct 16. PMID 24140548
- [Result] Di Stasi SM, Giannantoni A, Vespasiani G, Navarra P, Capelli G, Massoud R, Stephen RL. Intravesical electromotive administration of oxybutynin in patients with detrusor hyperreflexia unresponsive to standard anticholinergic regimens. J Urol. 2001 Feb;165(2):491-8. doi: 10.1097/00005392-200102000-00032. PMID 11176403
- [Result] Jost WH, Benecke R, Hauschke D, Jankovic J, Kanovsky P, Roggenkamper P, Simpson DM, Comella CL. Clinical and pharmacological properties of incobotulinumtoxinA and its use in neurological disorders. Drug Des Devel Ther. 2015 Apr 1;9:1913-26. doi: 10.2147/DDDT.S79193. eCollection 2015. PMID 25897202
- [Result] Veeratterapillay R, Harding C, Teo L, Vasdev N, Abroaf A, Dorkin TJ, Pickard RS, Hasan T, Thorpe AC. Discontinuation rates and inter-injection interval for repeated intravesical botulinum toxin type A injections for detrusor overactivity. Int J Urol. 2014 Feb;21(2):175-8. doi: 10.1111/iju.12205. Epub 2013 Jul 2. PMID 23819724
- [Result] Frevert J. Response to Commentary by W. Jost on: Pharmaceutical, Biological, and Clinical Properties of Botulinum Neurotoxin Type A Products. Drugs R D. 2015 Jun;15(2):217-8. doi: 10.1007/s40268-015-0091-y. No abstract available. PMID 25851380
- [Result] Benecke R. Clinical relevance of botulinum toxin immunogenicity. BioDrugs. 2012 Apr 1;26(2):e1-9. doi: 10.2165/11599840-000000000-00000. PMID 22385408
- [Result] Wang L, Sun Y, Yang W, Lindo P, Singh BR. Type A botulinum neurotoxin complex proteins differentially modulate host response of neuronal cells. Toxicon. 2014 May;82:52-60. doi: 10.1016/j.toxicon.2014.02.004. Epub 2014 Feb 21. PMID 24560879
- [Result] Jost WH, Blumel J, Grafe S. Botulinum neurotoxin type A free of complexing proteins (XEOMIN) in focal dystonia. Drugs. 2007;67(5):669-83. doi: 10.2165/00003495-200767050-00003. PMID 17385940
- [Result] Kumar R, Zhou Y, Ghosal K, Cai S, Singh BR. Anti-apoptotic activity of hemagglutinin-33 and botulinum neurotoxin and its implications to therapeutic and countermeasure issues. Biochem Biophys Res Commun. 2012 Jan 13;417(2):726-31. doi: 10.1016/j.bbrc.2011.12.020. Epub 2011 Dec 11. PMID 22182409
- [Result] Campanati A, Giuliodori K, Martina E, Giuliano A, Ganzetti G, Offidani A. Onabotulinumtoxin type A (Botox((R))) versus Incobotulinumtoxin type A (Xeomin((R))) in the treatment of focal idiopathic palmar hyperhidrosis: results of a comparative double-blind clinical trial. J Neural Transm (Vienna). 2014 Jan;121(1):21-6. doi: 10.1007/s00702-013-1074-1. Epub 2013 Sep 20. PMID 24052109